CLINICAL TRIAL: NCT06786065
Title: A Path to Prevention of Elder Abuse in Long-term Care. General Population Prevalence Study
Acronym: APPEAL
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other); City of Gothenburg (Unknown); Karolinska Institutet (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Johanna Simmons, Principal investigator, Linkoeping University
Other Study IDs: 2023-07931-01; A Path to Prevention of Elder (Other Grant/Funding Number: FORTE - Swedish Research Council for health, working life and welfare.)
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Elder Abuse
Keywords: Abuse of older people
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
The goal of this cross-sectional study is to learn about how common experiences of different forms of abuse are among people over the age of 65 years in Sweden. The main question it aims to answer is:

• What is the prevalence of abuse of older people in Sweden?

Participants are recruited through a random selection of people over 65 years from the populations register. Eligible participants are asked to answer a questionnaire including items about experiences of emotional, physical, sexual or financial abuse as well as neglect.

DETAILED DESCRIPTION:
Detailed Description Main aim

- Investigate the prevalence of abuse of older people in Sweden

Secondary aims:

* Investigate factors associated with reporting abusive experiences, e.g., health factors, frailty, care dependence
* Investigate resilience factors associated with abusive experiences, e.g., social support, positive emotion regulation and sense of purpose.

Study design and data collection Cross-sectional questionnaire study using a combination of digital and postal questionnaires and carried out by Statistics Sweden. A national representative sample of older adults will be used.

The invitation to participate and questionnaire will be sent to altogether 16 000 older adults (≥ 65 years) selected from the population register at random. To be able to provide information about experiences of abuse among both men and women, in all age groups and among the most vulnerable population, older adults residing in care facilities, the sample is stratified according to the information given in the study population description. Population weights will be used in analyses.

Material:

The questions about abusive experiences used in the study is part of the "REAGERA-S20" questionnaire developed and validated in a separate study (Clinical Trial register number NCT06659822). In addition, other relevant and validated questionnaires are included, e.g., The Tilburg Frailty Indicator, the UCLA loneliness scale, the Positive Emotional Regulation scale and a scale measuring sense of purpose.

In addition, statistics from Swedish registers concerning e.g., usage of home care services, sociodemographic factors and indicators of health status will be used to explore factors associated with elder abuse on different levels of the socio-ecological framework.

Analysis:

Prevalence will be reported for the different types of abuse (emotional, physical, sexual, financial abuse and neglect) in different relational contexts (partner, child, staff, other known perpetrator, unknown perpetrator).

Regression analyses will be used to investigate associations between reporting different forms of abuse and factors on different levels of the socio-ecological model. On an individual and relational level characteristic of respondents, e.g., age, educational level, own previous victimization, resilience factors as well as frailty and different health indicators from registers will be considered. On the community and societal level factors such as living conditions will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older (born in 1959 or earlier)

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Random sample (n=16 000) of adults age 65 or older from the Swedish population register. Sample is stratified in the following way:
  Age 65-74 years - 2000 men and 2000 women Age 75-84 years - 2000 men and 2000 women Age >85 years - 2000 men and women Registerd as living in an assissted living facility, age 65 or older - 2000 men and women
Sampling Method: Probability Sample
Enrollment: 7727 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of emotional abuse of older people | Day1. Cross sectional study using only one point of data collection. Participants are enrolled by returing a questionnaire including items about abuse. The timeframe used in the questionnaire is experiences of abuse during the past 12 months.
  Prevalence of emotional abuse the past 12 months as reported in part two of the REAGERA-S20 (Responding to Elder Abuse in Geriatric care) questionnaire. The questionnaire include five questions about emotional abusive experiences and each question is answered with yes or no. Yes to at least one question will be considered as reporting experiences of emotional abuse.
Prevalence of physical abuse of older people | Day 1. Cross sectional study using only one point of data collection. Participants are enrolled by returing a questionnaire including items about abuse. The timeframe used in the questionnaire is experiences of abuse during the past 12 months.
  Prevalence of physical abuse the past 12 months as reported in part two of the REAGERA-S20 (Responding to Elder Abuse in Geriatric care) questionnaire. The questionnaire include two questions about physical abusive experiences and each question is answered with yes or no. Yes to at least one question will be considered as reporting experiences of physical abuse.
Prevalence of sexual abuse of older people | Day 1. Cross sectional study using only one point of data collection. Participants are enrolled by returing a questionnaire including items about abuse. The timeframe used in the questionnaire is experiences of abuse during the past 12 months.
  Prevalence of sexual abuse the past 12 months as reported in part two of the REAGERA-S20 (Responding to Elder Abuse in Geriatric care) questionnaire. The questionnaire include two questions about sexually abusive experiences and each question is answered with yes or no. Yes to at least one question will be considered as reporting experiences of sexual abuse.
Prevalence of financial abuse of older people | Day 1. Cross sectional study using only one point of data collection. Participants are enrolled by returing a questionnaire including items about abuse. The timeframe used in the questionnaire is experiences of abuse during the past 12 months.
  Prevalence of financial abuse the past 12 months as reported in part two of the REAGERA-S20 (Responding to Elder Abuse in Geriatric care) questionnaire. The questionnaire include one questions about financial abusive experiences and is answered with yes or no. Yes to will be considered as reporting experiences of financial abuse.
Prevalence of neglect of older people | Day 1. Cross sectional study using only one point of data collection. Participants are enrolled by returing a questionnaire including items about abuse. The timeframe used in the questionnaire is experiences of abuse during the past 12 months.
  Prevalence of neglect the past 12 months as reported in part two of the REAGERA-S20 (Responding to Elder Abuse in Geriatric care) questionnaire. The questionnaire include two questions about neglect and each question is answered with yes or no. Yes to at least one question will be considered as reporting experiences of neglect.
Life-course prevalence of emotional abuse | Day 1
  Prevalence of emotional abuse over the life-course as reported in the questionnaire used. One question is used and possible answeres are "no", "yes before the age of 18", "yes between 18 and 65 years" and "yes after the age of 65 years". Results will be reported for abusive experience in each age span.
Life-course prevalence of physical abuse | Day 1
  Prevalence of physical abuse over the life-course as reported in the questionnaire used. One question is used and possible answeres are "no", "yes before the age of 18", "yes between 18 and 65 years" and "yes after the age of 65 years". Results will be reported for abusive experience in each age span.
Life-course prevalence of sexual abuse | Day 1
  Prevalence of sexual abuse over the life-course as reported in the questionnaire used. One question is used and possible answeres are "no", "yes before the age of 18", "yes between 18 and 65 years" and "yes after the age of 65 years". Results will be reported for abusive experience in each age span.
Life-course prevalence of financial abuse | Day 1
  Prevalence of financial abuse over the life-course as reported in the questionnaire used. One question is used and possible answeres are "no", "yes before the age of 18", "yes between 18 and 65 years" and "yes after the age of 65 years". Results will be reported for abusive experience in each age span.
Life-course prevalence of neglect | Day 1
  Prevalence of neglect over the life-course as reported in the questionnaire used. One question is used and possible answeres are "no", "yes before the age of 18", "yes between 18 and 65 years" and "yes after the age of 65 years". Results will be reported for abusive experience in each age span.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Simm, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linkoeping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be made available from the researcher upon reasonable request.